CLINICAL TRIAL: NCT05216939
Title: Assessment of Cloth Face Coverings as Source Control Under Laboratory and Simulated Field Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Colleen S. Kraft, Professor of Medicine, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY00001556
Record Dates: First submitted 2021-11-23; First posted 2022-02-01 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Masks

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Flannel mask with earl loops (Experimental): Participants will wear a flannel mask with earl loops
  Interventions: Other: Flannel mask with ear loops
- Flannel mask with ties (Experimental): Participants will wear a flannel mask with earl ties
  Interventions: Other: Flannel mask with ties
- Twill mask with ear loops (Experimental): Participants will wear a twill mask with ear loops
  Interventions: Other: Twill mask with ear loops
- Twill mask with ties (Experimental): Participants will wear a twill mask with ties
  Interventions: Other: Twill mask with ties

INTERVENTIONS:
Other: Flannel mask with ear loops — Participants will have a mask fit test and will wear a flannel mask with ear loops. While wearing the flannel mask, participants will perform a sequence of activities. The researchers will note whether the mask lost its fit (e.g., slipping off the nose or face). Between activities, participants will be told to re-adjust the mask. Participants will be assigned to a specific speed on a treadmill with no incline, either 1.5 mph, the 'light' activity level, or 3 mph, the 'moderate' activity level. They will walk on the treadmill for 10 minutes. Prior to the treadmill activity, participants will rate the comfort and fit of the mask. Near the end of the activity, participants will rate their perceived exertion and again rate the comfort of the mask. Participants will complete a post-experiment questionnaire following all activities.
  Arms: Flannel mask with earl loops
Other: Flannel mask with ties — Participants will have a mask fit test and will wear a flannel mask with ties. While wearing the flannel mask, participants will perform a sequence of activities. The researchers will note whether the mask lost its fit (e.g., slipping off the nose or face). Between activities, participants will be told to re-adjust the mask. Participants will be assigned to a specific speed on a treadmill with no incline, either 1.5 mph, the 'light' activity level, or 3 mph, the 'moderate' activity level. They will walk on the treadmill for 10 minutes. Prior to the treadmill activity, participants will rate the comfort of the mask. Near the end of the activity, participants will rate their perceived exertion and again rate the comfort of the mask. Participants will complete a post-experiment questionnaire following all activities.
  Arms: Flannel mask with ties
Other: Twill mask with ear loops — Participants will have a mask fit test and will wear a twill mask with ear loops. While wearing the twill mask with ear loops, participants will perform a sequence of activities. The researchers will note whether the mask lost its fit (e.g., slipping off the nose or face). Between activities, participants will be told to re-adjust the mask. Participants will be assigned to a specific speed on a treadmill with no incline, either 1.5 mph, the 'light' activity level, or 3 mph, the 'moderate' activity level. They will walk on the treadmill for 10 minutes. Prior to the treadmill activity, participants will rate the comfort of the mask. Near the end of the activity, participants will rate their perceived exertion and again rate the comfort of the mask. Participants will complete a post-experiment questionnaire following all activities.
  Arms: Twill mask with ear loops
Other: Twill mask with ties — Participants will have a mask fit test and will wear a twill mask with ties. While wearing the twill mask with ties, participants will perform a sequence of activities. The researchers will note whether the mask lost its fit (e.g., slipping off the nose or face). Between activities, participants will be told to re-adjust the mask. Participants will be assigned to a specific speed on a treadmill with no incline, either 1.5 mph, the 'light' activity level, or 3 mph, the 'moderate' activity level. They will walk on the treadmill for 10 minutes. Prior to the treadmill activity, participants will rate the comfort of the mask. Near the end of the activity, participants will rate their perceived exertion and again rate the comfort of the mask. Participants will complete a post-experiment questionnaire following all activities.
  Arms: Twill mask with ties

SUMMARY:
Cloth masks have been evaluated as a potential substitute for personal protective equipment (PPE) and found lacking. Prior to the COVID-19 outbreak, the use of cloth masks was limited and the focus of the limited research available was on the filtration of various fabrics in comparison to either surgical masks or N95 respirators. The Centers for Disease Control and Prevention (CDC) guidance for the coronavirus (COVID-19) outbreak makes it clear that cloth masks are not to be considered as PPE for healthcare workers and should be used in the healthcare setting only as a last resort when no other masks or respirators are available. While cloth masks are not recommended to be used as PPE, the use of cloth masks as primary source control has not yet been examined.

DETAILED DESCRIPTION:
This study will recruit children ages 6-11 and adults ages 18-65 living in the Atlanta/Metro-Atlanta area.

Participants will be randomly assigned to wear one of four different masks. These masks are created by combining one of two different kinds of fabric (flannel or twill) and one of two attachment devices (elastic ear loops or fabric ties). Additionally, adult participants will be randomly assigned to wear the mask while walking on a treadmill at either 1.5 mph or 3.0 mph. While wearing each mask, participants will perform the following sequence of activities: In a normal standing position, participants will 1) breathe normally (without talking), 2) breathe slowly and deeply, taking caution so as not to hyperventilate, 3) slowly turn his/her head from side to side between the extreme positions on each side, 4) slowly move his/her head up and down, inhaling in the up position (i.e., when looking toward the ceiling), 5) count up from 0-20 loudly and slowly, 6) grimace by smiling or frowning, 7) bend at the waist as if he/she were to touch his/her toes, and 8) breathe normally (without talking). Each activity will be performed for 1 minute, except for the grimace exercise, which will be performed for 15 seconds.

During the first two activities, the researcher will hold a mirror at each edge of the mask (nose, cheeks, and chin) to monitor whether there is fogging on the mirror. For the rest of the exercises, the researchers will note whether the mask lost its fit (e.g., slipping off the nose or face). Between activities, participants will be told to re-adjust the mask.

In the second phase of research activities, participants will walk on a treadmill while wearing their randomly assigned mask. Adult participants will be assigned to a specific speed on the treadmill with no incline, either 1.5 mph, the 'light' activity level, or 3 mph, the 'moderate' activity level. Child participants will only walk at 1.5 mph. Participants will walk on the treadmill for 10 minutes. Prior to the treadmill activity, the researcher will clip a probe to the participant's ear lobe that will measure transcutaneous carbon dioxide (CO2) (i.e., non-invasively) and pulse rate continuously during the performance of all physical activities. Prior to the treadmill activity, participants will rate the comfort of the mask. Near the end of the activity, participants will their perceived exertion and again rate the comfort of the mask. During the activity, participants will be free to adjust their masks as often as needed to maintain comfort and fit. The researcher will tally the frequency at which each participant adjusts their mask and the number of times that the mask lost its fit (e.g., slipping off the nose or face) and was not adjusted. Participants will complete a post-experiment questionnaire following all activities.

ELIGIBILITY:
Inclusion Criteria:

* Children between the ages of 6-11 years old
* Adults aged 18-65
* Adults who have never smoked or have smoked less than 100 cigarettes in their lifetime

Exclusion Criteria:

* Adults unable to consent
* Pregnant women
* Prisoners
* Cognitively impaired or Individuals with Impaired Decision-Making Capacity
* Individuals who are not able to clearly understand English
* Our research team does not have the resources required to translate our study materials or provide a translator for the study visit
* Any known cardiorespiratory condition (including but not limited to asthma, bronchitis, cystic fibrosis, congenital heart disease, and emphysema)
* Any known medical conditions that can be exacerbated by physical exercise (including but not limited to exercise-induced asthma, lower respiratory infections in the past 2 weeks, diabetes, hypertension, or epilepsy/seizure disorders)
* Any physical disability from a medical, orthopedic, or neuromuscular disorder that would interfere with the performance of physical activities
* Adult participants who are current or former smokers (i.e., an adult who has smoked 100 cigarettes in their lifetime and who currently smoke cigarettes, or an adult who has smoked 100 or more cigarettes in their lifetime)
* Inability to move the head from side to side or bend at the waist
* Inability to walk on a treadmill unassisted for the study duration
* Inability to tolerate wearing a mask while completing physical activities
* Anyone with symptoms of COVID-19 in the two weeks before their study visit
* Presence of an acute upper respiratory tract infection or symptomatic rhinitis (i.e., blocked nasal passages, runny nose, or significant sneezing) on the day of the study

Ages: 6 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2021-11-08 (Actual); Primary Completion 2022-02-22 (Actual); Study Completion 2022-02-22 (Actual)

PRIMARY OUTCOMES:
Change in Effect of masks textile types and designs on user discomfort | Before treadmill and after treadmill use (15 minutes)
  In order to better understand the effectiveness of different cloth masks for source control, the research team will assess the usability of the optimal masks through simulations by measuring comfort by using the optimal combinations of head suspension and mask designs. Participants will rate the discomfort of the mask they come in wearing and then rate the discomfort of the test mask they wear during the study after walking on a treadmill. Participants will answer the Discomfort of Cloth Masks-12 (DCM-12) scale which is comprised of 12 questions. For each item, there are four choices that correspond to four levels of discomfort: 1 (not at all), 2 (a little bit), 3 (somewhat), 4 (very much so). Items 1, 2, 4, 8, 10, and 12 will be used to obtain a subscale-score for breathability-related discomfort. Items 3, 5, 6, 7, 9, and 11 will be used to obtain a subscale-score for tightness-related discomfort. A higher score reflects a higher discomfort.
Change in the Effect of masks textile types and designs on their ability to stay in place. | Before and during treadmill use (from start up to 10 minutes)
  In order to better understand the effectiveness of different cloth masks for source control, the research team will assess the usability of the optimal masks through simulations by measuring the ability of the mask to stay in place. The research team will use a tally during the treadmill activity across the following: Touching face (no mask), touching mask (but no removing), Removed mask (remind to put back on).

SECONDARY OUTCOMES:
Change in heart rate | During treadmill: from start up to 10 minutes
  Prior to the treadmill activity, the researcher will clip a pulse rate continuously during the performance of all physical activities. Participants will walk on the treadmill for 10 minutes at either 1.5 or 3 miles per hour while wearing the assigned mask.
Monitoring of oxygen levels | During treadmill: from start up to 10 minutes
  Participants wearing the assigned mask will walk on the treadmill at either 1.5 or 3 miles per hour while their oxygen levels are monitored using a transcutaneous monitor.
Monitoring levels of carbon dioxide | During treadmill: from start up to 10 minutes
  Participants wearing the assigned mask will walk on the treadmill at either 1.5 or 3 miles per hour while their CO2 levels are monitored using a transcutaneous monitor.
Change in perceptions of mask comfort | Baseline (Before treadmill use) and immediately after treadmill up to 10 minutes
  Survey data on perceived exertion after fit mask test before treadmill use and after treadmill use

CONTACTS AND LOCATIONS:
Overall Officials: Colleen Kraft, MD, MSc, Principal Investigator — Emory University; Andrea L Shane, MD MPH MSc, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Emory Children's Center, Atlanta, Georgia
  - Emory University, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: Yes
The research team will share Individual participant data that underlie the results reported in the article, after deidentification.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: The research team will share data Immediately following the publication and ending 36 months following publication.
Access Criteria: All proposals should be directed to jmmumma@emory.edu. To gain access, data requestors will need to sign a data access agreement